CLINICAL TRIAL: NCT00321074
Title: AN OPEN, MULTICENTRE, RANDOMISED PARALLEL GROUP CLINICAL STUDY TO COMPARE SAFETY AND EFFICACY OF TACROLIMUS (FK506) WITH MONOCLONAL ANTI-IL2R ANTIBODIES (DACLIZUMAB) VS TACROLIMUS (FK506) WITH STEROIDS AND EVALUATE PHARMACOKINETICS IN LIVER ALLOGRAFT RECIPIENTS RECEIVING SUBOPTIMAL LIVERS
Brief Title: Tacrolimus and Daclizumab Versus Tacrolimus and Steroids in Liver Recipients Receiving Sub-optimal Grafts
Acronym: PANTERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-01-IT-02
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: LIVER TRANSPLANTATION
Keywords: IMMUNOSUPPRESSION; TACROLIMUS; MARGINAL LIVERS; PHARMACOKINETICS
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: TACROLIMUS
- 2 (Experimental)
  Interventions: Drug: TACROLIMUS

INTERVENTIONS:
Drug: TACROLIMUS — Immunosuppression
  Other Names: Prograf, FK506

SUMMARY:
The purpose of the study is to compare the safety and efficacy of two different tacrolimus based immunosuppressive regimens, one in combination with daclizumab, the other in combination with steroids, in recipients of suboptimal livers.

Pharmacokinetics of tacrolimus and bile composition will be measured in a subgroup of patients.

DETAILED DESCRIPTION:
Open, multicentre, 1:1 randomised, parallel group phase III study to compare safety and efficacy of tacrolimus (FK506) with monoclonal anti-IL2R antibodies (daclizumab) vs tacrolimus (FK506) with steroids and evaluate pharmacokinetics in liver allograft recipients receiving suboptimal livers.

Patients receiving primary suboptimal liver allograft transplantation (from donors > 65 years and/or liver macrosteatosis >15%) will be randomised to one of the following treatment arms:

Group I: steroid bolus (intraoperative) monoclonal anti-IL2R antibodies (daclizumab) induction tacrolimus Group II: steroid bolus (intraoperative) tacrolimus steroids

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Adult patients scheduled to receive a liver transplant
* Donors older than 65 and/or has liver macrosteatosis >15%
* Female patients of childbearing potential agree to maintain effective birth control during the study and must have negative pregnancy test at baseline

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than liver, or a liver re-transplantation.
* Patient has significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, or active peptic ulcer
* Patient is receiving an auxiliary graft or a bio-artificial liver has been used.
* Any pathology or medical condition that can interfere with this protocol study proposal
* Other exclusion applies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2005-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Incidence of and time to first biopsy-proven and treatment requiring acute rejection | 3 months

SECONDARY OUTCOMES:
Incidence of acute rejection | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (7):
- Italy (7):
  - Bergamo
  - Bologna
  - Milan
  - Padua
  - Roma
  - Torino
  - Udine

REFERENCES:
- See also: Link to FDA website — http://www.accessdata.fda.gov/scripts/cder/drugsatfda